CLINICAL TRIAL: NCT07258628
Title: Magnesium and Fentanyl in Preventing Reflex Hemodynamic Response to Endotracheal Intubation in Patients Aged 50 Years and Older
Brief Title: Comparison of Fentanyl and Magnesium to Control Reflex Hemodynamics in Patients Aged 50 and Older
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TABED 1-25-1089
Record Dates: First submitted 2025-09-19; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-09

CONDITIONS: Hypertension; Tachycardia
Keywords: Hemodynamic response; Elderly patients / age 50 and older; Magnesium sulfate; Fentanyl; Endotracheal intubation; Tachycardia; Hypertension
MeSH Terms: conditions — Hypertension; Tachycardia | interventions — Magnesium Sulfate; Solutions; Fentanyl

STUDY DESIGN:
Intervention Model Description: Single-center, three-arm, randomized, parallel-group interventional trial. Participants are assigned in a 1:1:1 ratio via sealed opaque envelopes to receive MgSO₄ 30 mg/kg IV over 10 minutes, MgSO₄ 30 mg/kg IV over 10 minutes plus fentanyl 2 mcg/kg IV, or fentanyl 2 mcg/kg IV. Masking: single-blind (outcome assessor/statistician); treating anesthesiologist is open-label. Standardized induction is performed with BIS and TOF monitoring; cases with laryngoscopy time >20 seconds are excluded. Primary endpoints are MAP and heart rate changes at baseline, post-intubation, and at 1-15 minutes after intubation.
Who Masked: Outcomes Assessor
Masking Description: In this trial, the anesthesiologist administering the study drugs is not blinded to group allocation. However, statistical analyses will be performed by an independent researcher who is blinded to treatment assignment. Therefore, the outcomes assessor is blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Magnesium Sulfate Infusion Group (30 mg/kg) (Experimental): Arm M: Magnesium sulfate (30 mg/kg IV over 10 min)
  Interventions: Drug: magnesium sulfate
- Fentanyl Only Group (2 mcg/kg) (Experimental): Participants will receive fentanyl 2 mcg/kg intravenously as a bolus
  Interventions: Drug: Fentanyl (IV)
- Combined Magnesium Sulfate (30 mg/kg) and Fentanyl (2 mcg/kg) Group (Experimental): Participants will receive magnesium sulfate 30 mg/kg intravenously over 10 minutes combined with fentanyl 2 mcg/kg intravenously
  Interventions: Drug: magnesium sulfate; Drug: Fentanyl (IV)

INTERVENTIONS:
Drug: magnesium sulfate — Magnesium sulfate 30 mg/kg administered intravenously over 10 minutes
  Other Names: MgSO₄; Epsom Salt; Magnesium Sulphate 15% Solution
  Arms: Combined Magnesium Sulfate (30 mg/kg) and Fentanyl (2 mcg/kg) Group; Magnesium Sulfate Infusion Group (30 mg/kg)
Drug: Fentanyl (IV) — Fentanyl 2 mcg/kg administered intravenously as a bolus
  Other Names: Fentanyl Citrate; Sublimaze; Talinat; Fentanyl Injection
  Arms: Combined Magnesium Sulfate (30 mg/kg) and Fentanyl (2 mcg/kg) Group; Fentanyl Only Group (2 mcg/kg)

SUMMARY:
This prospective, randomized, controlled trial aims to evaluate the effects of magnesium sulfate and fentanyl on the hemodynamic response to endotracheal intubation in surgical patients aged 50 years and older. A total of 75 patients will be enrolled and randomized into three groups: magnesium sulfate alone, magnesium sulfate plus fentanyl, and fentanyl alone. The primary outcome measures are changes in mean arterial pressure (MAP) and heart rate before and after intubation. Secondary outcomes include BIS, SEF, ST, TOF recovery times, intraoperative hemodynamic stability, and perioperative complications.

DETAILED DESCRIPTION:
Endotracheal intubation can trigger significant hemodynamic changes, such as tachycardia and hypertension, due to sympathetic activation. These responses are particularly detrimental in older patients with cardiovascular comorbidities, increasing the risk of perioperative morbidity and mortality.

The aim of this study is to compare the effectiveness of magnesium sulfate and fentanyl, administered alone or in combination, in attenuating the hemodynamic response to intubation in patients aged 50 years and older undergoing elective surgery.

This is a single-center, prospective, randomized, controlled trial. A total of 75 patients will be randomized into three groups:

Group M: Magnesium sulfate 30 mg/kg IV infusion over 10 minutes Group X: Magnesium sulfate 30 mg/kg IV infusion over 10 minutes plus fentanyl 2 mcg/kg IV Group F: Fentanyl 2 mcg/kg IV Standardized anesthesia induction and monitoring will be performed. The primary outcome measures are mean arterial pressure (MAP) and heart rate, recorded at baseline, post-induction, and at 1, 3, 5, 10, and 15 minutes after intubation. Secondary outcomes include BIS, SEF, and ST values; TOF recovery times; anesthesia duration; intraoperative blood loss; fluids and blood products administered; and perioperative complications.

The findings of this study are expected to provide valuable insights into the pharmacological management of intubation-induced hemodynamic responses in the elderly surgical population.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years
* Patients scheduled for elective surgery under general anesthesia
* Patients requiring endotracheal intubation with a single-lumen tube
* Provision of written informed consent

Exclusion Criteria:

* Known renal or hepatic insufficiency
* Thyroid dysfunction
* Uncontrolled hypertension
* Suspected difficult airway (Mallampati ≥ 3 or history of difficult intubation)
* Known allergy or hypersensitivity to study medications
* Myocardial infarction within the past 3 months
* Presence of heart block
* Preoperative hypermagnesemia

Withdrawal Criteria:

* Laryngoscopy time exceeding 20 seconds
* Withdrawal of informed consent
* Patient withdrawal from the study at any time

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2026-01-10 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Mean Arterial Pressure (MAP) Changes | Baseline (pre-induction), immediately after induction, and at 1, 3, 5, 10, and 15 minutes after intubation.
  Change in mean arterial pressure (MAP) to assess the hemodynamic response to endotracheal intubation. MAP will be measured at baseline (pre-induction), immediately after induction, and at 1, 3, 5, 10, and 15 minutes after intubation.
1. Heart Rate (HR) Changes | Baseline (pre-induction), immediately after induction, and at 1, 3, 5, 10, and 15 minutes after intubation.
  Change in heart rate to assess the hemodynamic response to endotracheal intubation. Heart rate will be measured at baseline (pre-induction), immediately after induction, and at 1, 3, 5, 10, and 15 minutes after intubation.

SECONDARY OUTCOMES:
Train of Four (TOF) Recovery Time | Intraoperatively when TOF count reaches 2.
  Time required for early neuromuscular recovery following administration of rocuronium. Continuous neuromuscular monitoring will be performed, and the duration from rocuronium injection until return of TOF count to 2 will be recorded.
Perioperative Complications | From immediately after endotracheal intubation up to 15 minutes post-intubation.
  Incidence of perioperative complications, including hypotension, hypertension, bradycardia, tachycardia, and arrhythmia, recorded during the first 15 minutes after endotracheal intubation.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Ankara Bilkent City Hospital, Department of Anesthesiology and Reanimation, Ankara
  - Ankara City Hospital, Ankara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Misganaw A, Sitote M, Jemal S, Melese E, Hune M, Seyoum F, Sema A, Bimrew D. Comparison of intravenous magnesium sulphate and lidocaine for attenuation of cardiovascular response to laryngoscopy and endotracheal intubation in elective surgical patients at Zewditu Memorial Hospital Addis Ababa, Ethiopia. PLoS One. 2021 Jun 1;16(6):e0252465. doi: 10.1371/journal.pone.0252465. eCollection 2021. PMID 34061894
- [Background] Aissaoui Y, Qamous Y, Serghini I, Zoubir M, Salim JL, Boughalem M. Magnesium sulphate: an adjuvant to tracheal intubation without muscle relaxation--a randomised study. Eur J Anaesthesiol. 2012 Aug;29(8):391-7. doi: 10.1097/EJA.0b013e328355cf35. PMID 22717726
- [Background] James MF, Beer RE, Esser JD. Intravenous magnesium sulfate inhibits catecholamine release associated with tracheal intubation. Anesth Analg. 1989 Jun;68(6):772-6. PMID 2735543